CLINICAL TRIAL: NCT03692923
Title: Impact of A Peer Virtual Community on Pregnant Women's Well-being: A Quasi-experimental Study
Brief Title: VIRTUAL COMMUNITY for PREGNANT WOMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, WAN-RU WU, Assistant Professor, Tzu Chi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TCU
Record Dates: First submitted 2018-09-21; First posted 2018-10-02 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Normal Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): participants received ordinary prenatal care.
- virtual community group (Experimental): participants were invited to join a virtual community to interact with peers in addition to their ordinary prenatal care.
  Interventions: Other: virtual community

INTERVENTIONS:
Other: virtual community
  Arms: virtual community group

SUMMARY:
The study aimed to investigate the effect of exclusive peer-to-peer virtual support on pregnant women's well-being including physical symptoms, depression, social support, maternal attachment, and pregnancy adaptation.

DETAILED DESCRIPTION:
The pregnancy period is marked by not only the joy and excitement of bonding with her baby but also dramatic changes in her body. The Internet's convenience and anonymity provide great possibilities for pregnant women to create a social network for sharing personal stories, seeking information and asking questions, and expressing own emotions and concerns.

Although health-related online communities are emerging rapidly around the globe, little is known about the impact of a virtual peer community on pregnant women's well-being.

The study enrolled 138 pregnant women, who were assigned to either the experimental or control groups. After obtaining informed consent from participants, we asked them to fill out the baseline questionnaires (Time 1). The first and second follow-ups (Times 2 and 3) were conducted at 22-24 and 36-38 weeks of pregnancy, respectively. Participants in the experimental group received ordinary prenatal care in addition to virtual community participation, and those in the control group received only ordinary prenatal care.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women were older than 20 years old
2. Had at least 9 years of education.

Exclusion Criteria:

1. Had complications in this pregnancy
2. Had underlying medical problems with pregnancy.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
The pregnancy adaptation scale | repeated measured at second trimester (22-24 weeks of pregnancy), and the third trimester (36-38 weeks of pregnancy).
  Used to investigate the changes in the scores of pregnancy adaptation. Items are scored from 0 to 3 and they are summed to compute a total score ranging from 0 to 84. Higher scores indicate better pregnancy adaptation.
The Edinburgh Depression Scale | repeated measured at second trimester (22-24 weeks of pregnancy), and the third trimester (36-38 weeks of pregnancy).
  Used to investigate the changes in the scores of depression. Items are scored from 0 to 3 and they are summed to compute a total score ranging from 0 to 30. The cut-off point for depression is a total score of 12 or above.

SECONDARY OUTCOMES:
The Symptoms Checklist | repeated measured at second trimester (22-24 weeks of pregnancy), and the third trimester (36-38 weeks of pregnancy).
  Used to investigate the changes in the scores of pregnancy-related physical symptoms. Items are scored from 1 to 4 and they are summed to compute a total score ranging from 22 to 88. Higher scores indicate experiencing more symptoms.
The Social Support Scale | repeated measured at second trimester (22-24 weeks of pregnancy), and the third trimester (36-38 weeks of pregnancy).
  Used to investigate the changes in the scores of social support perception. Items are scored from 1 to 5 and they are summed to compute a total score ranging from 20 to 100. higher scores indicate perceived higher social support from family, peer pregnant women, friends, and healthcare providers.
The Maternal-Fetal Attachment Assessment Scale | repeated measured at second trimester (22-24 weeks of pregnancy), and the third trimester (36-38 weeks of pregnancy).
  Used to investigate the changes in the scores of maternal-fetal attachment. Items are scored from 1 to 5 and they are summed to compute a total score ranging from 39 to 195. Higher scores indicate higher maternal-fetal attachment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu WR, Hung CH. Impact of a peer virtual community on pregnant women's well-being: A repeated-measure and quasi-experimental study. J Adv Nurs. 2019 May;75(5):1099-1107. doi: 10.1111/jan.13938. Epub 2019 Jan 24. PMID 30575093